CLINICAL TRIAL: NCT06495450
Title: PROVE-VR: A Pilot Randomized Trial Using Omnidirectional Virtual Reality and Treadmill Training for Chronic Stroke Survivors
Brief Title: Using Omnidirectional Virtual Reality and Treadmill Training for Chronic Stroke
Acronym: PROVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Brain Canada (Other)
Responsible Party: Principal Investigator, Adria Quigley, Assistant Professor, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PROVE_stroke
Record Dates: First submitted 2024-06-20; First posted 2024-07-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Stroke
Keywords: Virtual Reality; Stroke rehabilitation; Omnidirectional treadmill
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omni-VR group (Experimental): 20 participants will undergo 45-minute training sessions 3 times per week for 12 weeks using omnidirectional virtual reality and treadmill training.
  Interventions: Device: Omnidirectional Virtual Reality and Treadmill Training
- Control group (Active Comparator): 10 participants will undergo 45-minute traditional physiotherapy training sessions including lower limb strengthening and unidirectional treadmill training 3 times per week for 12 weeks.
  Interventions: Behavioral: Traditional Exercise

INTERVENTIONS:
Device: Omnidirectional Virtual Reality and Treadmill Training — Omni-VR forest scenario developed by our team involving real-life dual task walking and dynamic balance activities (ie. stepping over obstacles, and managing distractions) will be used for treatment group.
  Arms: Omni-VR group
Behavioral: Traditional Exercise — A traditional exercise program including strengthening and unidirectional treadmill activities for the same duration will be completed in control group.
  Arms: Control group

SUMMARY:
The primary objective of this pilot randomized controlled trial (RCT) is to test the feasibility (consent rate, retention rate, participant burden, adherence, technical issues, safety) and usability (system usability scale, SUS) of Omnidirectional treadmill Virtual Reality training (omni-VR) among chronic stroke survivors. Our secondary objective is to (1) estimate the extent to which cognition, brain activation during a dual task activity, walking ability, and dynamic balance change after 3 months of training among intervention participants (omni-VR) and traditional exercise controls, and (2) estimate the extent to which health-related quality of life and motivation co-evolve with our secondary outcomes.

Researchers will compare the intervention group and control group to evaluate the impact of omni-VR on cognition and physical function among stroke survivors.

Participants will:

* undergo a 45-minute training session 3 times per week for 12 weeks
* intervention group: omni-VR
* control group: traditional exercise program (strengthening and walking activities)

DETAILED DESCRIPTION:
Mounting data indicates that cognition plays a role in complex walking and balance. However, conventional intervention methods lack a sufficient incentive to encourage participants to adhere to the treatment. Further, it is difficult to provide a substantial amount of treatment to induce cortical reorganization.

Virtual reality or VR (a computer-generated simulation of 3-dimensional virtual environments that reacts in real time to the user's actions) has been introduced to neurorehabilitation to promote improvements in walking ability, balance, and cognition. It has also been demonstrated to be effective in improving motivation among stroke survivors and augmenting neuroplasticity.

Omnidirectional treadmill technology can be integrated with VR to allow for fully immersive rehabilitation. This novel and innovative technology mimics real-world environments and maximizes challenging cognitive and physical dual-tasking and balance activities while maintaining patient safety. However, no randomized trials have evaluated the impact of omnidirectional treadmill VR (Omni-VR) on cognitive and physical function among stroke survivors.

Therefore, our study aims to test the feasibility and usability of the Omni-VR. This pilot randomized control trial will also be the first study to test the feasibility and effect of a fully-immersive active omni-VR system among chronic stroke survivors

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18
* Stroke ≥ 6 months ago (confirmed with chart review)
* Living within 50 km of Halifax, Nova Scotia
* Functional Ambulation Category of 3 or greater on a scale of 0-5, to ensure the participant is able to walk with supervision or independently. This criterion was selected to ensure participants could safely participate in the intervention.
* Ability to participate in low-moderate intensity aerobic or strengthening exercise for ≥ 15 minutes to ensure participants can tolerate intervention sessions of 30-45 minutes, with activity breaks, in keeping with previous stroke rehabilitation studies.
* No uncorrected visual deficits or spatial neglect
* No cardiovascular, orthopedic, or neurological diseases other than stroke impacting walking or balance
* Can follow simple instructions
* Score of < 27 on the adapted Motion Sickness Susceptibility Scale-Short based on established normative values indicating more than moderate susceptibility to motion sickness.

Exclusion Criteria:

* Unstable serious medical condition
* Resting blood pressure >180/100mmHg
* History of abnormal untreated heart rhythm
* Pregnancy
* Condition limiting ability to complete or tolerate the exercises without major program modifications (e.g., chronic low back pain)
* Serious comorbid condition that would affect participation in the intervention (e.g., active cancer, severe heart disease)
* Severe loss of hearing or speech that would preclude VR use
* Participant weight more than 264 lbs (weight limit for Virtualizer Elite 2 treadmill)
* Participating in another formal lower limb exercise program > 1 day per week
* History of QT prolongation or using potential QT prolonging drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-09-06 (Estimated)

PRIMARY OUTCOMES:
Consent rate | Baseline
  Consent rate is the percentage of eligible individuals who participate. The investigators expect a consent rate of at least 40%.
Retention rate | 12 weeks (study completion)
  Retention rate is the percentage of participants who complete the 12-week intervention. The investigators expect a retention rate of 80% for the intervention group.
Usability of the Omnidirectional Treadmill and Virtual Reality Game | 12 weeks (study completion)
  Usability will be assessed by System Usability Scale (SUS) out of 100 points. The investigators expect a SUS score of 71 or higher among all participants.
Participant burden | Baseline and 12 weeks (study completion)
  Participant burden will be measured by the percentage of participants finishing assessments in 100 minutes or less. The investigators anticipate at least 85% of participants completing assessments within the time limit.
Adherence | 12 weeks (study completion)
  Adherence will be measured by the exercise session attendance. The investigators expect the treatment group to attend 70% or more of the sessions.
Equipment downtime | 12 weeks (study completion)
  The investigators will record any treadmill downtime due to VR technical issues. The targets are zero significant downtime in 85% of sessions.
Equipment safety | 12 weeks (study completion)
  The investigators will record any serious adverse events related to the study. The target is no serious adverse events related to the study

SECONDARY OUTCOMES:
Cognitive function | Baseline and 12 weeks (study completion)
  The investigators will use the Computerized MoCA [Montreal Cognitive Assessment] Duo to evaluate participants' cognitive function.
Executive Function | Baseline and 12 weeks (study completion)
  The investigators will use the Dimensional Change Card Sort to evaluate participants' executive function.
Working memory | Baseline and 12 weeks (study completion)
  The investigators will use the List Sorting Working Memory Test to evaluate participants' working memory.
Brain activation in prefrontal and premotor cortices | Baseline and 12 weeks (study completion)
  Brain activation using fNIRS [Functional near-infrared spectroscopy] in the prefrontal and premotor regions of interest during a single task (steady-state omnidirectional treadmill walking) and two cognitive-physical dual-task activities (simple dual-task: steady-state omnidirectional treadmill walking while repeating the same word and complex dual-task: steady-state omnidirectional treadmill walking while performing a verbal fluency test)
Walking Speed | Baseline and 12 weeks (study completion)
  Walking speed using VIVE trackers on omnidirectional treadmill and overground
Step cadence | Baseline and 12 weeks (study completion)
  The investigators will evaluate step cadence using the VIVE trackers.
Step width | Baseline and 12 weeks (study completion)
  The investigators will evaluate step width using the VIVE trackers.
Step length | Baseline and 12 weeks (study completion)
  The investigators will evaluate step length using the VIVE trackers.
Dynamic balance | Baseline and 12 weeks (study completion)
  The investigators will measure the static sway with feet together using omni-VR system and use MINI-BESTest to measure the dynamic balance.

OTHER OUTCOMES:
Motivation of participant | 12 weeks (study completion)
  The investigators will measure motivation by intrinsic motivation inventory. Higher scores indicate better results.
Health-related quality of life of participant | Baseline and 12 weeks (study completion)
  The investigators will measure health-related quality of life by the Stroke Impact Scale-3.0. Higher scores indicate better results.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Rehabilitation & Arthritis Centre, Halifax, Nova Scotia, Canada